CLINICAL TRIAL: NCT04586556
Title: Artificial Intelligence for Real-time Detection and Monitoring of Colorectal Polyps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 20.198
Record Dates: First submitted 2020-10-01; First posted 2020-10-14 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Adenomatous Polyps
Keywords: Polyps detection; Artificial Intelligence; Adenoma detection; Polyps classification; Quality indicators
MeSH Terms: conditions — Adenomatous Polyps

STUDY DESIGN:
Intervention Model Description: prospective, multi-endoscopist, single center, clinical study at tertiary referral center (CHUM)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Artificial intelligence for real-time detection and monitoring of colorectal polyps (Experimental): A standard colonoscopy will be performed according to the standard of routine care. All optically diagnosed polyps will be removed and sent to the CHUM pathology laboratory for histopathological evaluation according to institutional standards. The AI system will capture video of the procedure in real time, and provide additional information on the detection of polyps, follow-up and prediction of pathology. The full-length colonoscopy videos will be annotated for the exact time of the identification of the anatomical landmarks, polyps, also for polyp- and procedural-related characteristics.
  Interventions: Diagnostic Test: Polyps detection by Artificial Intelligence

INTERVENTIONS:
Diagnostic Test: Polyps detection by Artificial Intelligence — The AI system will capture the live video of the procedure and the AI feedback (polyp detection, tracking, and pathology prediction) will be shown on a second screen installed next to the regular endoscopy screen. Screen A will show the regular endoscopy image and screen B will show the regular endoscopy image together with the areas that might harbor a polyp or the information to predict pathology

SUMMARY:
The investigators hypothesize that the clinical implementation of a deep learning AI system is an optimal tool to monitor, audit and improve the detection and classification of polyps and other anatomical landmarks during colonoscopy. The objectives of this study are to generate preliminary data to evaluate the effectiveness of AI-assisted colonoscopy on: a) the rate of detection of adenomas; b) the automatic detection of the anatomical landmarks (i.e., ileocecal valve and appendiceal orifice).

DETAILED DESCRIPTION:
In this trial, the investigators aim to evaluate the followings:

1. the accuracy of automatic detection of important anatomical landmarks (i.e., ileocecal valve, appendiceal orifice);
2. the accuracy of automatic detection of polyps/adenomas (PDR/ADR);

ELIGIBILITY:
Inclusion Criteria :

* Signed informed consent
* Age 45-80 years
* Indication to undergo a lower GI endoscopy.

Exclusion Criteria :

* Coagulopathy
* Poor general health, defined as an American Society of Anesthesiologists (ASA) physical status class >3
* Emergency colonoscopies
* Hospitalized patients
* Known inflammatory bowel disease (IBD)
* Patients currently in the emergency room

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 372 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-05-11 (Actual)

PRIMARY OUTCOMES:
Number of polyps detected | Day 1
  Efficacy of AI assisted colonoscopy to detect the proportion of patients with at least 1 polyp. Polyp detection rate with an AI.
Evaluation of the automatic report of the colonoscopy quality indicators | Day 1
  Compare of the automatic detection of the ileocecal valve, appendiceal orifice, and the automatic calculation of the withdrawal time with manual detection

CONTACTS AND LOCATIONS:
Overall Officials: Daniel von Renteln, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (3):
- Canada (2):
  - Université de Montréal, Montreal, Quebec
  - Centre Hospitalier Universitaire de Montréal, Montreal, Quebec
- IHU Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No